CLINICAL TRIAL: NCT00208494
Title: Comparative Study to Evaluate the Safety and Efficacy of the DePuy Ceramic-on-metal Total Hip Prosthesis Versus the DePuy Metal-on-metal Total Hip Prosthesis Through Clinical and Radiographical Data
Brief Title: Metal on Metal Versus Ceramic on Metal Hip Replacement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: DePuy Orthopaedics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 03062
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Results first posted 2011-08-04 (Estimated); Last update posted 2013-08-14 (Estimated); Status verified 2013-08

CONDITIONS: Non-inflammatory Joint Diseases
Keywords: Non-Inflammatory Degenerative Joint Disease
MeSH Terms: interventions — Arthroplasty, Replacement, Hip

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Active Comparator): Ceramic-on-metal total hip implant
  Interventions: Device: Total Hip Replacement
- B (Active Comparator): Metal-on-metal total hip implant
  Interventions: Device: Total hip replacement

INTERVENTIONS:
Device: Total Hip Replacement — Total hip replacement
  Other Names: Biolox Delta head; Ultamet insert; Pinnacle Acetabular shell
  Arms: A
Device: Total hip replacement — Total hip replacement
  Other Names: CoCr M-head, Ultamet insert, Pinnacle Acetabular shell
  Arms: B

SUMMARY:
The purpose of this study is to compare the performance of artificial hips with metal heads and metal sockets to artificial hips with ceramic heads articulating with metal socket components. The success of the total hip arthroplasty (THA) will be based upon all of the following clinical and radiographic criteria being met at the two-year evaluation: (1) the patient's clinical results as measured using modified Harris Hip evaluation rating system, and the absence of a complication that requires the surgical removal or replacement of a component; and (2) radiographic findings at study endpoint (i.e., two years follow-up). Clinical and radiographic success at two (2) years postoperative is required for the study hip to be deemed successful.

DETAILED DESCRIPTION:
This study is a prospective, multi-center, randomized, single blind, controlled clinical investigation comparing the safety and efficacy of the cementless Ceramic on Metal total hip prostheses versus the cementless Metal on Metal total hip prostheses.

ELIGIBILITY:
Inclusion Criteria:

* Able to (or capable of) provide consent to participate in the clinical investigation prior to the day of the surgery.
* Skeletally mature (tibial and femoral epiphyses are closed)
* Undergoing cementless primary hip replacement surgery for Noninflammatory Degenerative Joint Disease
* Affected hip has a Harris Hip Score of 70 or lower and a Pain rating of Moderate or greater
* Radiographic Parameters:
* X-Ray Evaluation confirms the presence of NIDJD
* Femoral and acetabular bone stock is sufficient, regarding strength and shape, and is suitable to receive the implants
* No structural bone grafts required to support to prosthetic component(s)or to shape the bone to receive implant(s)
* Willing to have knowledge of treatment arm (CoM or MoM) withheld for a period of 24 months post-operatively unless disclosure is legally and/or medically necessary
* Previous THA in contralateral hip that is greater than one (1) year postoperative and has a Harris Hip pain rating less than MILD

Exclusion Criteria:

* Bilateral hip disease with the anticipated need for bilateral hip implant during study participation (i.e., within the next 24 months)
* THA required for the revision of a previously failed THA
* Suffering from inflammatory arthritis
* Prior prosthetic hip replacement
* Previous Girdlestone procedure or surgical fusion in the operative hip joint
* Above knee amputation of either the contralateral or ipsilateral leg
* Known allergy to metal (e.g. jewelry)
* The presence of highly communicable disease or diseases that may limit follow-up (e.g., immuno-compromised conditions, hepatitis, active tuberculosis, etc.)
* Significant neurological or musculoskeletal disorders or disease that may adversely affect gait or weight bearing (e.g., muscular dystrophy, multiple sclerosis)
* Conditions that may interfere with the total hip arthroplasty survival or outcome (e.g., Paget's disease, Charcot's disease)
* Unwilling or unable to comply with a rehabilitation program for a cementless THA or difficulty or inability to return for follow-up visits prescribed by the study protocol
* Known to be pregnant, a prisoner, mentally incompetent, and/or alcohol or drug abuser
* Previous treatment for renal disease
* Any systemic steroid therapy, excluding inhalers, within three months prior to surgery

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 392 (Actual)
Dates: Start 2005-08; Primary Completion 2008-12 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Scott, MD, Principal Investigator — Orthopaedic Specialty Clinic; Patrick G Kirk, MD, Principal Investigator; Shekhar S Desai, MD, Principal Investigator; Charles A Engh, Jr., MD, Principal Investigator — Anderson Clinic; Ajai Cadambi, MD, Principal Investigator — Adult Orthopaedic Reconstruction Texas Hip and Knee Center; C L Barnes, MD, Principal Investigator — Foundation for Musculoskeletal Research & Education
Locations (9):
- United States (8):
  - Foundation for Musculoskeletal Research and Education, Little Rock, Arkansas
  - Orange, California
  - Palm Bay, Florida
  - Charlotte, North Carolina
  - Cincinnati, Ohio
  - Anderson Clinic, Alexandria, Virginia
  - Roanoke, Virginia
  - Spokane, Washington
- London, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eleven sites enrolled 392 subjects who were then randomized into two groups. The investigational group, Ceramic-on-Metal (COM) and the control group, Metal-on-Metal (MOM). Two subjects were intraoperatively excluded, resulting in 194 subjects COM subjects and 196 MOM subjects.
Groups:
- Ceramic-on-Metal (COM) Total Hip Implant: The COM modular total hip prosthesis has a ceramic femoral head articulating with a metal alloy acetabular bearing insert.
- Metal-on-Metal (MOM) Total Hip Implant: The MOM modular total hip prosthesis has a metal femoral head articulating with a metal alloy acetabular bearing insert.
Period: Overall Study
Arm/Group | Ceramic-on-Metal (COM) Total Hip Implant | Metal-on-Metal (MOM) Total Hip Implant
Started | 194 | 196
Completed | 164 | 162
Not Completed | 30 | 34

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ceramic-on-Metal (COM) Total Hip Implant | Metal-on-Metal (MOM) Total Hip Implant | Total
Number analyzed (Participants) | 194 | 196 | 390
Age Continuous [Mean (Standard Deviation); unit: Years]
  Age | 58.9 (10.1) | 59.1 (9.5) | 59 (9.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 83 | 91 | 174
  Male | 111 | 105 | 216
Region of Enrollment [Number; unit: participants]
  United States | 194 | 196 | 390

OUTCOME MEASURES:

1. Primary Outcome: Composite Success/Failure
Description: The composite success/failure of the implant was made up of radiographic, clinical and revision data. Radiographic success was determined by femoral subsidence =/< 2mm, acetabular migration =/< 2mm, cup inclination =/< 4°, no acetabular or femoral osteolysis, and acetabular and femoral lucencies less than 50% of visible porous coating. Clinical success was determined by a Harris Hip score equal to or greater than 80. A hip (patient) was considered to be a composite success at study endpoint if it was a radiographic and clinical success and no revision of any component had taken place.
Time Frame: At 24 months
Population: Out of the 390 subjects, 84 subjects were removed from the analysis for the following reasons: 2 deaths (1 in each arm); 3 protocol violations (2 COM, 1 MOM); 28 bilateral (12 COM, 16 MOM); 39 subjects had no 24-month Harris Hip score (22 COM, 17 MOM); and 12 subjects had no 24-month x-ray (4 COM, 8 MOM).
Measure: Number; unit: Participants
Arm/Group | Ceramic-on-Metal (COM) Total Hip Implant | Metal-on-Metal (MOM) Total Hip Implant
Number analyzed (Participants) | 154 | 152
Participants | 142 | 141

ADVERSE EVENTS:
Arm/Group | Ceramic-on-Metal (COM) Total Hip Implant | Metal-on-Metal (MOM) Total Hip Implant
Serious Adverse Events (participants affected / at risk) | 40/194 | 48/196
Other Adverse Events (participants affected / at risk) | 137/194 | 125/196
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ceramic-on-Metal (COM) Total Hip Implant (N=194) | Metal-on-Metal (MOM) Total Hip Implant (N=196)
Bone Fracture (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 2 (2)
Cardiovascular (Cardiac disorders) | 5 (5) | 4 (4)
Central Nervous System (Nervous system disorders) | 3 (3) | 2 (2)
Constitutional Symptom (General disorders) | 0 (0) | 1 (1)
Dermatological (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dislocation (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Gastrointestinal (Gastrointestinal disorders) | 5 (5) | 2 (2)
Genitourinary (Renal and urinary disorders) | 3 (3) | 1 (1)
Hematological (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
Hematoma requiring drainage (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 21 (21) | 23 (23)
Operative Adverse Event (fracture of femur (Surgical and medical procedures) | 3 (3) | 8 (8)
Operative Adverse Event (other complication (Surgical and medical procedures) | 0 (0) | 2 (2)
Operative Adverse Event (seating acetabular prosthesis) (Surgical and medical procedures) | 0 (0) | 2 (3)
Peripheral nervous system (Nervous system disorders) | 0 (0) | 1 (1)
Respiratory system (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Deep Infection (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ceramic-on-Metal (COM) Total Hip Implant (N=194) | Metal-on-Metal (MOM) Total Hip Implant (N=196)
Trochanteric Bursitis (Musculoskeletal and connective tissue disorders) | 15 (15) | 10 (10)
Central Nervous System (Nervous system disorders) | 14 (14) | 14 (14)
Genitourinary (Renal and urinary disorders) | 15 (15) | 19 (19)
Respiratory system (Respiratory, thoracic and mediastinal disorders) | 16 (16) | 19 (19)
Dermatological (Skin and subcutaneous tissue disorders) | 31 (31) | 24 (24)
Hematological (Blood and lymphatic system disorders) | 14 (14) | 17 (17)
Cardiovascular (Cardiac disorders) | 25 (25) | 20 (20)
Gastrointestinal (Gastrointestinal disorders) | 19 (19) | 19 (19)
Constitutional symptom (General disorders) | 21 (21) | 17 (17)
Wound problem (Injury, poisoning and procedural complications) | 12 (12) | 11 (11)
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 106 (106) | 91 (91)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less